CLINICAL TRIAL: NCT03648723
Title: The Comparison of the Effect of Periodontal Treatment in Patients With Diabetic and Non Diabetic Nephropathy
Brief Title: The Effect of Periodontal Disease Treatment in Patients With Kidney Disease
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Zekeriya Tasdemir, Principal investigator, TC Erciyes University
Other Study IDs: Ztasdemir
Record Dates: First submitted 2018-08-22; First posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic nephropathy: Diabetic nephropathy is defined by macroalbuminuria that is, a urinary albumin excretion of more than 300 mg in a 24-hour collection or macroalbuminuria and abnormal renal function as represented by an abnormality in serum creatinine, or glomerular filtration rate(GFR)
- Non-diabetic nephropathy: This group consisted of diagnosis with nephropathy without diabetes mellitus.

SUMMARY:
the purpose of the present study was to compare the effects of non-surgical periodontal therapy by clinical and biochemical parameters on patients undergoing continous ambulatory peritoneal dialysis(CAPD) due to diabetic nephropathy and non-diabetic

DETAILED DESCRIPTION:
A new branch of periodontology, deﬁned as "medical periodontology," has been proposed that mentioned the bidirectional relationship between periodontal disease and systemic conditions.

In the lights of these informations, the purpose of the present study was to compare the effects of non-surgical periodontal therapy on patients undergoing continous ambulatory peritoneal dialysis(CAPD) due to diabetic nephropathy and non-diabetic. Forty three participants ( 22 Diabetic Nephropathy(DN) group , 21 Non-Diabetic Nephropathy(N-DN) group) were included and divided into the two group; DN group and N-DN group, in the present study.

The following clinical parameters were evaluated at baseline and the end of the study: Plaque index ; Gingival index ; pocket depth (PD) measurements; bleeding on probing (BOP)-percentage of BOP (+) sites; gingival recession (GR)-from the cement-enamel junction to the gingival margin; and clinical attachment level (CAL)-the sum of PD and GR measurements. The Decay-Missing-Filling Index (DMFT) was recorded. Clinical examinations were repeated 6 months following periodontal treatment. All clinical measurements were taken from the mid-buccal and mid-lingual sites and the buccal aspects of the interproximal contact area for the mesial and distal sites of each tooth to the nearest 0.5 mm using a 15 mm periodontal probe at baseline and the 6th months after treatment. All periodontal clinical examinations were performed by one calibrated examiner (FOT). At baseline and 6 months after treatment, fasting venous blood samples were collected from the antecubital fossa by an experienced nurse. Blood samples for TNF- α, IL-6 and PTX-3 were centrifuged, and separated serum and plasma samples were stored at -80◦C until analysis. TNF-α , IL-6 , and PTX-3 serum levels were determined using a commercial solid-phase enzyme-linked immunosorbent assay (ELISA) kit according to the manufacturer's instructions. Periodontal treatments were performed 2 hours after the patients had their breakfast following the blood sampling. Standard oral hygiene instructions were given to all groups, including interdental plaque control (interdental brushes) and brushing of the dorsum of the tongue twice a day. Oral hygiene control and re-instructions were provided during all visits. After local infiltration, full-mouth scaling and root planning (FM-SRP) was performed by the same investigator with standard periodontal curettes

ELIGIBILITY:
Inclusion Criteria:

* had to have chronic periodontitis
* ≥15 natural teeth
* needed to be >30 years old

Exclusion Criteria:

* History of antibiotic or anti-inflammatory drugs within the previous 6 months
* pregnancy or lactation
* periodontal therapy within 6 months prior to the study
* past or current smoking and alcohol consumption

Ages: 31 Years to 65 Years
Age Groups: Adult, Older Adult
Study Population: All patients in each groups had to have chronic periodontitis and ≥15 natural teeth; moreover, they needed to be >30 years old. History of antibiotic or anti-inflammatory drugs within the previous 6 months, pregnancy or lactation, periodontal therapy within 6 months prior to the study, past or current smoking and alcohol consumption were considered to be exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2016-01-10 (Actual); Primary Completion 2017-01-10 (Actual); Study Completion 2017-05-10 (Actual)

PRIMARY OUTCOMES:
Periodontal disease parameters change | Examinations were performed at baseline and repeated 6 months following periodontal treatment. Change is determined with at baseline - at 6 months after periodontal treatment.
  pocket depth (mm) evaluation .was performed by periodontal probe.

SECONDARY OUTCOMES:
Biochemical parameters change | biochemical parameters were evaluated at baseline and 6 months following periodontal treatment . Change is determined with baseline - 6 months after periodontal treatment.
  TNF-α pg/mL serum levels were evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Zekeriya Taşdemir, Principal Investigator — TC Erciyes University

IPD SHARING:
Plan to Share IPD: Undecided